CLINICAL TRIAL: NCT00365053
Title: Phase II Study of PXD101 (NSC 726630) as Second-Line Therapy for Treatment of Patients With Malignant Pleural Mesothelioma
Brief Title: PXD101 as Second-Line Therapy in Treating Patients With Malignant Mesothelioma of the Chest That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02839; PHII 67; N01CM62209 (NIH)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Advanced Malignant Mesothelioma; Epithelial Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — belinostat

ARMS (1):
- Treatment (belinostat) (Experimental): Patients receive PXD101 IV at 1000 mg/m2 over 30 minutes on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: belinostat; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: belinostat — Given IV
  Other Names: PXD101
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well PXD101 works as second-line therapy in treating patients with malignant mesothelioma of the chest that cannot be removed by surgery. PXD101 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with unresectable malignant pleural mesothelioma (MPM) treated with PXD101.

SECONDARY OBJECTIVES:

I. Determine the overall survival and time to progression in these patients. II. Assess the toxicities associated with this drug in these patients. III. Perform molecular correlative studies on tumor tissue (optional) and peripheral blood (required) and identify potential predictive markers for response.

OUTLINE:

Patients receive PXD101 IV over 30 minutes on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection during course 1 of treatment for biomarker correlative studies. Fetal hemoglobin (hemoglobin F) levels are measured via reverse transcriptase-polymerase chain reaction as a potential predictive marker for response.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant pleural mesothelioma (MPM) of any of the following subtypes:

  * Epithelial
  * Sarcomatoid
  * Mixed
* Have received only 1 prior systemic chemotherapy regimen for advanced mesothelioma

  * Prior intrapleural cytotoxic agents (including bleomycin) not considered systemic chemotherapy
  * Patients who are not candidates for combination chemotherapy are eligible even if they have not received prior chemotherapy
* Unresectable disease
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan

  * The sole site of measurable disease must not be located within the radiotherapy port
* No known brain metastases
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* WBC >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin normal
* AST/ALT =< 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance >= 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception for 1 week before, during, and for >= 2 weeks after completion of study treatment
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to PXD101
* No symptomatic congestive heart failure
* No congestive heart failure related to primary cardiac disease
* No unstable angina pectoris
* No cardiac arrhythmia
* No condition requiring anti-arrhythmic therapy
* No uncontrolled hypertension
* No myocardial infarction within the past 6 months
* No ischemic or severe valvular heart disease
* No ongoing or active infection
* No marked baseline prolongation of QT/QTc interval
* No repeated QTc interval > 500 msec
* No long QT syndrome
* No other significant cardiovascular disease
* No other uncontrolled intercurrent illness
* No psychiatric illness or social situation that would preclude study compliance
* Recovered from prior therapy
* No prior valproic acid or other known histone deacetylase (HDAC) inhibitor
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 3 weeks since prior radiation therapy
* No concurrent medication that may cause torsade de pointes
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Belinostat)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 73 [27 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate According to the Response Evaluation Criteria in Solid Tumors (RECIST) Committee
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT, MRI or X-ray: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 13
percentage of participants | 0

2. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 13
Months | 4.5 [2.3 to 5.3]

3. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 3 years
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 13
Months | 1.2 [1.1 to 1.6]

4. Secondary Outcome: Toxicity Profile
Description: Toxicity information recorded will include the type, severity, time of onset, time of resolution, and the probable association with the study regimen. Toxicities table summarizes the observed incidence by severity and type of toxicity for toxicities that are related to treatment and greater than grade 1. Adverse events assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 13
Participants
  Grade 2 : Hemoglobin | 6
  Grade 2 : Lymphopenia | 1
  Grade 2 : Albumin | 1
  Grade 2 : Anorexia | 2
  Grade 2 : AST | 0
  Grade 2 : Constipation | 2
  Grade 2 : Creatinine | 1
  Grade 2 : Sweating | 1
  Grade 2 : Dyspnea | 3
  Grade 2 : Fatigue | 0
  Grade 2 : Glucose (hyperglycemia) | 6
  Grade 2 : Hypoxia | 0
  Grade 2 : Hypotension | 1
  Grade 2 : Infection | 2
  Grade 2 : Nausea | 2
  Grade 2 : Pain | 1
  Grade 2 : Sodium (Hyponatremia) | 0
  Grade 2 : Supraventricular arrhythmia NOS | 2
  Grade 3 : Hemoglobin | 0
  Grade 3 : Lymphopenia | 0
  Grade 3 : Albumin | 0
  Grade 3 : Anorexia | 0
  Grade 3 : AST | 1
  Grade 3 : Constipation | 0
  Grade 3 : Creatinine | 0
  Grade 3 : Sweating | 0
  Grade 3 : Dyspnea | 1
  Grade 3 : Fatigue | 2
  Grade 3 : Glucose (hyperglycemia) | 0
  Grade 3 : Hypoxia | 0
  Grade 3 : Hypotension | 0
  Grade 3 : Infection | 0
  Grade 3 : Nausea | 0
  Grade 3 : Pain | 0
  Grade 3 : Sodium (Hyponatremia) | 3
  Grade 3 : Supraventricular arrhythmia NOS | 1
  Grade 4 : Hemoglobin | 0
  Grade 4 : Lymphopenia | 0
  Grade 4 : Albumin | 0
  Grade 4 : Anorexia | 0
  Grade 4 : AST | 0
  Grade 4 : Constipation | 0
  Grade 4 : Creatinine | 0
  Grade 4 : Sweating | 0
  Grade 4 : Dyspnea | 1
  Grade 4 : Fatigue | 0
  Grade 4 : Glucose (hyperglycemia) | 0
  Grade 4 : Hypoxia | 1
  Grade 4 : Hypotension | 0
  Grade 4 : Infection | 0
  Grade 4 : Nausea | 0
  Grade 4 : Pain | 0
  Grade 4 : Sodium (Hyponatremia) | 0
  Grade 4 : Supraventricular arrhythmia NOS | 0

5. Secondary Outcome: Apoptosis by TUNEL Assay
Description: Summarized with contingency tables or scatterplots, and with quantitative measures of agreement.
Time Frame: At baseline
Population: Assay data were not collected.
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 0

6. Secondary Outcome: Histone Acetylation by IHC and Western Blotting
Description: Summarized with contingency tables or scatterplots, and with quantitative measures of agreement.
Time Frame: At baseline and at 4 hours after last dose of PXD101 on day 5
Population: IHC data were not collected.
Arm/Group | Treatment (Belinostat)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 1 year, 1 month.
Description: "Other" adverse events table includes all grades and attributions to treatment not included in the "Serious" adverse events table.
Arm/Group | Treatment (Belinostat)
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Belinostat) (N=13)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Belinostat) (N=13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 8 (11)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 8 (13)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 10 (15)
Vomiting (Gastrointestinal disorders) | 7 (9)
Chest pain (General disorders) | 3 (4)
Disease progression (General disorders) | 9 (9)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 10 (16)
Fever (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Hypersensitivity (Immune system disorders) | 2 (2)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3)
Alkaline phosphatase increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Creatinine increased (Investigations) | 4 (4)
Haptoglobin decreased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (3)
Lymphopenia (Investigations) | 1 (1)
Weight loss (Investigations) | 5 (8)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 3 (7)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (9)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (19)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 3 (5)
Hypertension (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Phlebitis superficial (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less